CLINICAL TRIAL: NCT01403090
Title: A Single Treatment, Open Label, Multicenter, Safety Study of the Angel™ Catheter in Hospitalized Human Subjects With a Temporary Risk of Pulmonary Embolism
Brief Title: Safety Study of the Angel™ Catheter in Subjects With Risk of Pulmonary Embolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BiO2 Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CPR-001
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Venous Thromboembolism
Keywords: Pulmonary Embolism; Deep Vein Thrombosis; Venous Thromboembolism; Central Line Catheter; Vena Cava Filters
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Angel Catheter (Experimental)
  Interventions: Device: Angel Catheter

INTERVENTIONS:
Device: Angel Catheter — The Angel Catheter will be inserted in the femoral vein following standard central line placement techniques. Once the catheter is on the Inferior Vena Cava, the filter will be deployed following the manufacturer instructions and secured to the skin.

SUMMARY:
The Angel™ Catheter combines the functions of a vena cava filter and a multi-lumen central line catheter. The device is designed to be placed in the inferior vena cava via the femoral vein for the prevention of Pulmonary Embolism (PE) and for access to the central venous system. The primary endpoint is freedom from serious adverse events (SAE), defined as death, symptomatic pulmonary embolism or major bleeding .

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years and older
2. Be admitted to the hospital

   One of the following two criteria:
3. Patients with proven deep vein thrombosis (DVT) or pulmonary embolism ( PE), at high risk for pulmonary embolism and under consideration for insertion of a retrievable inferior vena cava (IVC) filter with at least one of the following criteria:

   * Contraindications for anticoagulation
   * Recurrent PE despite adequate anticoagulation
   * Emergency treatment following massive pulmonary embolism
4. Patients at high risk for developing PE who require but have a temporary or absolute contraindication for prophylaxis with anticoagulation, including:

   * Patients with multiple trauma and active or recent bleeding with contraindications to anticoagulation or that require a temporary stop of anticoagulation
   * severe head injury with coma
   * severe hemorrhagic stroke with coma
   * head injury with a long bone fracture
   * spinal cord injury with paraplegia or quadriplegia
   * multiple (≥2) long bone fractures with pelvic fracture
   * multiple (≥4) long bone fractures
   * Critically ill patients in the Medical or Surgical Intensive Care Unit with high risk of PE that require but are contraindicated for anticoagulation prophylaxis and will benefit from a temporary filter and a central venous access catheter
   * Patients who had recently undergone or are about to undergo a surgical procedure that requires temporary interruption of anticoagulation for Venous Thromboembolism (VTE) and will benefit from a temporary vena cava filter and central

Exclusion Criteria:

1. Patient is less than 18 years
2. Patient is pregnant or has a positive serum human chorionic gonadotropin (HCG) pregnancy test at baseline visit
3. Patient or next legal representative cannot give informed consent
4. Patients with anticipated survival < 2 days (catastrophic illness)
5. Body mass index greater than 35
6. Patient has a pre-existing filter
7. Participation in another simultaneous interventional medical investigation or interventional trial.
8. Patient has indications for a permanent filter at the time of the initial evaluation
9. Patient has an uncontrollable coagulopathy with active bleeding.
10. Patient with proven endocarditis or bacteremia
11. Patient has hypersensitivity to any of the components of the Angel™ Catheter, specifically Nitinol
12. Known acute or chronic thrombotic occlusion of both common femoral veins or iliac veins
13. Patient with functioning pelvic renal allograft on the only side available for device insertion
14. Patient who will undergo surgical procedure involving the femoral vein or pelvic veins through which the device must be inserted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Cadavid, MD, Principal Investigator — Hospital Pablo Tobon Uribe; Bladimir Gil, MD, Principal Investigator — Clinica Las Americas
Locations (2):
- Colombia (2):
  - Clinica las Americas, Medellín, Antioquia
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started at the Hospital Pablo Tobon Uribe and was then followed at the clinical las Americas. Eight patients were recruited in the initial phase of the study
Groups:
- Angel Catheter: Angel Catheter Placement : The Angel Catheter will be inserted in the femoral vein following standard central line placement techniques. Once the catheter is on the Inferior Vena Cava, the filter will be deployed following the manufacturer instructions and secured to the skin.
Period: Overall Study
Arm/Group | Angel Catheter
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Angel Catheter
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.4 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  Colombia | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Device safety was evaluated on the basis of identification and summarization of the incidence rates of complications and adverse effects.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Angel Catheter
Number analyzed (Participants) | 8
participants | 0

ADVERSE EVENTS:
Arm/Group | Angel Catheter
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angel Catheter (N=8)
Death (Infections and infestations) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less